CLINICAL TRIAL: NCT06911424
Title: A Phase 3 Randomized, Multi-Center, Placebo-Controlled, Masked Study to Evaluate the Clinical Efficacy and Safety of Fusidic Acid 1% Viscous Topical Antibiotic Eye Drops for the Treatment of Suspected Bacterial Conjunctivitis
Brief Title: Efficacy of Fusidic Acid 1% in the Treatment of Bacterial Conjunctivitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Baxis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BXP-301
Record Dates: First submitted 2025-03-19; First posted 2025-04-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Bacterial Conjunctivitis
Keywords: Conjunctival Diseases; Eye Diseases; Eye Infections, Bacterial; Bacterial Infections; Infections; Eye Infections; Conjunctivitis, Bacterial; Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial; Conjunctival Diseases; Eye Diseases; Eye Infections, Bacterial; Bacterial Infections; Infections; Eye Infections; Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: All study staff (Sponsor, Site and Contract Research Organization (CRO)) involved in the day to day activities of the study are masked. Each site will have a designated unmasked dosing coordinator and the Sponsor/CRO will have an unmasked team member(s) as well, who is not involved in study conduct (e.g., for investigational product or statistical activities that require an unmasked individual).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fusidic Acid 1% (Experimental): Participants will instill one drop of fusidic acid 1% per eye twice a day (BID) for 7 days. Approximately 12 hours between doses is preferred, but BID administration takes precedence over precise timing
  Interventions: Drug: Fusidic Acid 1%
- Placebo (Placebo Comparator): Participants will instill one drop of Placebo ophthalmic solution per eye BID for 7 days. Approximately 12 hours between doses is preferred, but BID administration takes precedence over precise timing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fusidic Acid 1% — Fusidic acid 1%
  Arms: Fusidic Acid 1%
Drug: Placebo — Placebo ophthalmic solution
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to demonstrate the superiority of fusidic acid 1% over placebo in adults and children with confirmed bacterial conjunctivitis and to further establish the safety profile of fusidic acid 1% for topical ocular administration.

ELIGIBILITY:
Main Inclusion Criteria:

* Have a clinical diagnosis of suspected bacterial conjunctivitis in at least 1 eye, confirmed by the presence of purulent or mucopurulent ocular discharge and a grade ≥ 1 on the modified Validated Bulbar Redness (VBR) conjunctival redness scale.
* Have not received any ocular treatment for conjunctivitis, aside from eyelid hygiene, ≤14 days prior to Visit 1.
* Have a negative viral conjunctivitis test in both eyes.
* Agree to discontinue use of eye/eyelid cosmetics during study participation.
* Agree to discontinue use of contact lenses during study participation.
* Be willing and able to provide informed consent and comply with the study requirements.
* Not be currently pregnant or breastfeeding. If sexually active, agree to use approved contraception for the duration of the study.

Main Exclusion Criteria:

* Have signs and/or symptoms or a diagnosis of fungal, protozoal, or viral etiology ≤30 days prior to Visit 1.
* Have experienced signs and symptoms of bacterial conjunctivitis for >48 hours prior to Visit 1.
* Require or are expected to require use of any non-study topical ocular medication or systemic medications prior to Visit 1 as specified in the protocol as ineligible.
* Have any abnormality of the ocular anatomy or ocular disease/disorder specified in the protocol as ineligible.
* Have a known intolerance, sensitivity or allergy to the study medications or any of their components.
* Have participated in another clinical trial ≤30 days or received another experimental drug ≤90 days prior to Visit 1.
* Have a family member or household member enrolled in this study.
* Have a condition which in the investigator's opinion may impact their safety or would negatively affect the conduct or outcome of the study.
* Be an employee of or immediate family member of an employee (directly related to study conduct) at the study site.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Clinical Cure | Visit 2 (Day 4)
  Proportion of patients with a positive bacterial culture at Visit 1 (Day 1) who achieve clinical cure.

SECONDARY OUTCOMES:
Microbial Eradication | Visit 2 (Day 4)
  Proportion of subjects with a positive bacterial culture at Visit 1 (Day 1) who achieve microbiological eradication.
Microbial Eradication | Visit 3 (Day 8)
  Proportion of subjects with a positive bacterial culture at Visit 1 (Day 1) who achieve microbiological eradication.
Clinical Cure | Visit 3 (Day 8)
  Proportion of patients with a positive bacterial culture at Visit 1 (Day 1) who achieve clinical cure.

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Baxis Site 04, Little Rock, Arkansas
  - Baxis Site 24, Huntington Beach, California
  - Baxis Site 19, La Jolla, California
  - Baxis Site 39, Long Beach, California
  - Baxis Site 31, Los Angeles, California
  - Baxis Site 38, Los Angeles, California
  - Baxis Site 20, Sherman Oaks, California
  - Baxis Site 34, Delray Beach, Florida
  - Baxis Site 22, Doral, Florida
  - Baxis Site 11, Lake Worth, Florida
  - Baxis Site 37, Largo, Florida
  - Baxis Site 27, Lutz, Florida
  - Baxis Site 01, Miami, Florida
  - Baxis Site 03, Miami, Florida
  - Baxis Site 13, Miami Beach, Florida
  - Baxis Site 28, Miami Lakes, Florida
  - Baxis Site 29, Palm Springs, Florida
  - Baxis Site 10, Tampa, Florida
  - Baxis Site 35, Union City, Georgia
  - Baxis Site 15, Idaho Falls, Idaho
  - Baxis Site 06, Orland Park, Illinois
  - Baxis Site 26, Columbia, Maryland
  - Baxis Site 21, North Las Vegas, Nevada
  - Baxis Site 23, Babylon, New York
  - Baxis Site 05, Mount Airy, North Carolina
  - Baxis Site 25, Tulsa, Oklahoma
  - Baxis Site 30, Gresham, Oregon
  - Baxis Site 09, Pittsburgh, Pennsylvania
  - Baxis Site 12, Charleston, South Carolina
  - Baxis Site 33, Greenville, South Carolina
  - Baxis Site 08, Edinburg, Texas
  - Baxis Site 02, Humble, Texas
  - Baxis Site 14, Kingwood, Texas
  - Baxis Site 36, Mission, Texas
  - Baxis Site 17, Layton, Utah
  - Baxis Site 18, Layton, Utah
  - Baxis Site 16, West Valley City, Utah
  - Baxis Site 32, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No